CLINICAL TRIAL: NCT07048886
Title: Rocklatan Adds Pressure Reduction After MIGS (Minimally Invasive Glaucoma Surgery)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Center for Sight Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFS-RAPRAM-101; 96015755 (Other Grant/Funding Number: Alcon Vision, LLC)
Record Dates: First submitted 2025-06-15; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary Open Angle Glaucoma; Rocklatan
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — netarsudil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Comparator Systane Artificial Tears (Placebo Comparator): Comparator arm is Systane artificial tears
  Interventions: Drug: Systane
- FDA Approved Rocklatan (netarsudil 0.02% and latanoprost 0.005%) (Active Comparator): FDA approved Rocklatan (netarsudil 0.02% and latanoprost 0.005%) is a fixed dose combination of a Rho kinase inhibitor and a prostaglandin analogue indicated for the reduction of elevated intraocular pressure (IOP) in patients with open-angle glaucoma or ocular hypertension.
  Interventions: Drug: Rocklatan (netarsudil 0.02% and latanoprost 0.005%)

INTERVENTIONS:
Drug: Rocklatan (netarsudil 0.02% and latanoprost 0.005%) — Additional intraocular eye pressure lowering post-Hydrus
  Arms: FDA Approved Rocklatan (netarsudil 0.02% and latanoprost 0.005%)
Drug: Systane — Placebo Comparator (artificial tears)
  Arms: Placebo Comparator Systane Artificial Tears

SUMMARY:
The primary objective of this study is to determine if the addition of Rocklatan post-Hydrus will provide additional intraocular pressure lowering.

DETAILED DESCRIPTION:
The study is a prospective single-practice with multiple locations, single-surgeon, parallel double arm study in subjects with open angle glaucoma (OAG), who were implanted with Hydrus microstent combined with cataract surgery to be randomized to receive Rocklatan vs. Comparator (artificial tears). Unmedicated MDIOP (mean diurnal intraocular pressure) measurements will be assessed at baseline (after Hydrus, prior to study medication) and at 1-month post-initiation of Study Drop.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years and older
* Subjects who have mild to moderate Open Angle Glaucoma (OAG)
* Subjects who have undergone uncomplicated cataract surgery and Hydrus microstent implantation > 3 months prior to screening and within the last 2 years
* Post-Hydrus subjects on 0-2 ocular hypotensive medication classes who can safely washout (if on ocular hypotensive medications)
* Unmedicated or washed out IOP range between 16-26 mmHg

Exclusion Criteria:

* History of intraocular surgery except for uneventful refractive surgery or uncomplicated cataract surgery and hydrus microstent implantation
* Prior Selective Laser Trabeculoplasty (SLT) within 18 months of surgery
* Secondary glaucoma excluding pseudoexfoliation and pigmentary dispersion syndrome
* Severe Open Angle Glaucoma
* Narrow angles, other angle abnormalities or angle closure glaucoma
* Allergy or intolerance to Rocklatan
* History of corneal edema, or corneal disease or dystrophy
* Current or history of intra-ocular infection or inflammation
* History of retinal diseases that could affect diagnostic testing
* Anticipated use of intra-ocular or topical steroids not associated with the study protocol
* Pregnant, breastfeeding or planning to become pregnant during the study
* Any condition in the opinion in the investigator that would potentially confound the results of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean diurnal intraocular pressure change from baseline | After 28 days up to 35 days post initiation of Rocklatan vs placebo comparator
  After Hydrus prior to study initiation drop

SECONDARY OUTCOMES:
Diurnal Intraocular pressure change from baseline and difference between intraocular pressure at each time point | After Hydrus prior to study drop and after 28 days up to 35 days post initiation of study drop for all time points 8am, 10am, 4pm (± 1 hour) between groups
  Goldmann Applanation Tonometry

OTHER OUTCOMES:
Change in corneal hysteresis from baseline | Change from baseline after 28 days up to 35 days post initiation of study drop
  Ocular Response Analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Medical Doctor, Principal Investigator — Center For Sight
Locations (1):
- Center for Sight, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not plan to share individual participant data due to concerns about participant privacy and confidentiality.